CLINICAL TRIAL: NCT06541327
Title: Cellular Immunotherapy for Relapsed or Refractory Lymphoma Data Collection
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Other Study IDs: CCIC-001
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: CAR-T
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Receptors, Chimeric Antigen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAR-T: Chimeric antigen receptor modified T cells
  Interventions: Drug: Chimeric Antigen Receptor

INTERVENTIONS:
Drug: Chimeric Antigen Receptor — CAR-T
  Other Names: Chimeric antigen receptor modified T cells

SUMMARY:
This study aims to collect clinical data from adult patients with relapsed or refractory non-Hodgkin's lymphoma (r/r NHL) receiving cellular immunotherapy to establish a large database of cellular immunotherapy for Chinese patients.

DETAILED DESCRIPTION:
This study aims to collect efficacy and safety data from adult patients with r/r NHL who received cellular immunotherapy between January 2017 and December 2040. Study investigators will determine the most appropriate diagnostic and treatment plans for patients based on clinical practice, without any intervention due to the existence of this study. No grouping will be conducted, and subgroup analyses will be performed based on the collected data.

Data collection process:

Clinical data will be collected from patients before cellular immunotherapy, before immune cell infusion, on the day of infusion, and at the last visit or follow-up within 24 months post-infusion. This includes collecting efficacy data, adverse events related to cellular immunotherapy, and survival data. Additionally, any new tumors, pathological findings, and other relevant laboratory or auxiliary examination data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a confirmed diagnosis of r/r B-NHL (including r/r DLBCL, r/r FL, r/r MCL, HGBL-NOS, FL3b, r/r MZL, transformed lymphomas such as MCL) and r/r T-cell lymphoma, who have received informed consent waivers;
* Patients who have received or are receiving cellular immunotherapy, with cellular immunotherapy products including the following categories: cytokine-induced killer cell therapy (CIK), tumor-infiltrating lymphocytes (TIL), cytokine-induced killer cell-dendritic cell mixed therapy (DC-CIK), chimeric antigen receptor T cells, NK cells or macrophage therapy (CAR-T, CAR-NK, CAR-M), T-cell receptor chimeric T cell therapy (TCR-T), dendritic cell therapy.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsed or refractory lymphoma receiving cellular immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate in 3 months | 3 months post CAR-T infusion
  Complete Response rate in 3 months is defined as the incidence of subjects achieving complete remission (CR) within 3 months after CAR-T infusion according to the Lugano Classification (Cheson et al, 2014), as determined by study investigators.

SECONDARY OUTCOMES:
Objective remission rate (ORR) in 3months | 3 months post CAR-T infusion
  ORR in 3 moths is defined as the incidence of either a CR or a partial response (PR) within 3 months after CAR-T infusion per the Lugano Classification as determined by study investigators.
Overall Survival (OS) | 2 years post CAR-T infusion
  OS is defined as the time from CAR-T infusion to the date of death from any cause.
Adverse events (AEs) | 2 years post CAR-T infusion
  Types, frequency, and severity of adverse events and laboratory anomalies Physiological parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Shanghai Institute of Hematology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided